CLINICAL TRIAL: NCT03423290
Title: Safety and Efficacy Analysis of FRED™/FRED™Jr Embolic Device in Aneurysm Treatment, a UK, Multi-center, Single Arm, Prospective Observational Study
Brief Title: Safety and Efficacy Analysis of FRED™/FRED™Jr Embolic Device in Aneurysm Treatment
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Collaborators: Clinact (Other)
Responsible Party: Sponsor
Other Study IDs: FRED-UK Registry
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FRED and FRED Jr — Flow Re-Direction Endoluminal Device

SUMMARY:
A prospective, multicenter, observational evaluation of the safety and efficacy of the FRED® device in the treatment of intracranial aneurysms

DETAILED DESCRIPTION:
This is a multi-center observational study. Treatment and follow-up visits will be done as per standard of care.

The purpose of this study is to demonstrate that use of the FRED/FRED Jr Embolic device in intracranial aneurysm treatment is safe and effective when assessed at 1, 6 and 12 month post procedure.

100 patients will be enrolled over an 18-month recruitment period. All patients will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years old
2. Patient harboring an unruptured intracranial aneurysm:

   * for which endovascular treatment is indicated
   * for which use of FRED or FRED Jr has been deemed appropriate
   * being the only one to require treatment over the period of the study
   * and optionally previously treated by surgery (clipping) or with an intrasaccular device: aneurysm recanalized
3. Patient with a modified Rankin Scale (mRS) ≤ 2
4. Patient or patient's legally authorized representative has received information about data collection and has signed and dated an Informed Consent Form

Exclusion Criteria:

1. Patient has suffered an ICH within the 30 days prior to the procedure.
2. The aneurysm to be treated is associated with an cAVM
3. The aneurysm to be treated is a dissecting or blister-like aneurysm
4. The aneurysm to be treated or any other aneurysm is in the posterior circulation
5. The aneurysm to be treated has a stenosis of its parent artery
6. Patient has another aneurysm previously treated with a stent or a flow diverter

   * on the same parent vessel at any time (except in the case of the proximal carotid if the treatment occurred more than 3 months prior to the procedure)
   * on a different parent vessel, less than 3 months prior to the procedure
7. Patient has another aneurysm requiring treatment within the study period
8. Patient with a known allergy to antiplatelet, to heparin, to contrast products or nickel titanium
9. Patient with a contra-indication to antiplatelet or heparin
10. Pregnancy or child breastfeeding
11. Patient unable or unlikely to complete required follow up
12. Patient has severe or fatal comorbidity or a life expectancy of less than 1 year
13. Treatment with a flow diverter other than FRED/FRED Jr or in addition to FRED/FRED Jr is planned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged a minimum of 18 years with an unruptured or recanalized intracranial aneurysm in whom endovascular treatment has been determined the appropriate treatment
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Complete aneurysm occlusion without ˃ 50% parent artery stenosis | 6 months
  Evaluated by Corelab
Morbidity rate | 6 months
  patients with mRS>2
Mortality rate | 6 months
  patients with mRS=6

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Lobotesis, MD, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (7):
- United Kingdom (7):
  - University Hospital Birmingham, Birmingham
  - Brighton & Sussex Universitys Hospitals, Brighton
  - Western General Hospital - NHS Lothian, Edinburgh
  - The Walton Centre NHS Foundation Trust, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No